CLINICAL TRIAL: NCT07071064
Title: Mississippi Community Engagement Alliance (MS CEAL): Fostering Community Solutions
Acronym: MS CEAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Mississippi Food Network (Unknown); Mississippi State University (Other); Center for Family Life, Inc. (Unknown); Locust Grove MB Church (Unknown); Grace Episcopal Church (Unknown); Choctaw Health Center (Unknown)
Responsible Party: Principal Investigator, Caroline Compretta, Assistant Vice Chancellor for Research, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UMMC-IRB-2024-141; SUB-OTA No. 6922-03-COVID-S009 (Other Grant/Funding Number: NIH/Westat)
Record Dates: First submitted 2025-06-06; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Nutrition Security
Keywords: Nutrition Security; Health Literacy; Health Promotion; Community Engaged Research

STUDY DESIGN:
Intervention Model Description: In this study, individuals at each site will be randomly assigned to either the intervention group, which will receive the food boxes and nutrition education, or the control group, which will receive food boxes. Participants assigned to the control group will be offered the nutrition education program after data collection is complete. The project will employ simple randomization at a one-to-one basis as participants are randomized using random number generator. By measuring key process and clinical indicators before and after the intervention, the study team will assess the impact of the program on participants' nutritional status and overall health.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Food Box + Nutrition (Experimental): Participants receive a food box as well as nutrition classes
  Interventions: Behavioral: Food Box + Nutrition Classes
- Food Box (Active Comparator): Participants receive a food box only
  Interventions: Behavioral: Food Box Only

INTERVENTIONS:
Behavioral: Food Box + Nutrition Classes — The Nutrition Security Intervention is a 12-month project enrolling 400 adults across four sites. Participants will receive the intervention for 6 months, with a 9-month and 12-month in person follow-up. Individuals receiving this intervention will receive bi-weekly food boxes, containing 15-20 pounds of fresh produce, grains, and legumes. They will also participate in a bi-weekly nutrition class, led by a Registered Dietician.
  Arms: Food Box + Nutrition
Behavioral: Food Box Only — The intervention is a 12-month project enrolling 400 adults across four partner sites. Participants will receive the intervention for 6 months, with a 9-month and 12-month in person follow-up. In this intervention, participants will receive a bi-weekly food box only (no nutrition education) during the intervention period. They will have the opportunity to participate in the educational component after the completion of the intervention period.
  Arms: Food Box

SUMMARY:
The Mississippi Community Engagement Alliance (MS CEAL) Team proposes to address the complexities of Mississippi's health issues and social determinants of health through its Fostering Community Solutions (FOCUS) Project, with two objectives: (1) advance the health and wellbeing of Mississippi's populations experiencing differing health outcomes; and (2) enhance the resilience and power within communities to disseminate and implement evidence-based interventions. This study's specific aims include: (1) examine whether the inclusion of a nutrition education program increases fruit and vegetable consumption in a food box distribution program and (2) recruit and train community nutrition liaisons to implement sustainable community strategies to longitudinally support nutrition security. The primary outcome for the first specific aim will be fruit and vegetable consumption. Secondary outcome measures will include changes in perceptions and knowledge related to food consumption and dietary intake. Clinical outcomes will include changes in blood pressure, blood sugar, and cholesterol. For Specific Aim 2, outcomes will include the ability to recruit community nutrition liaisons at each site, the number of trainings, pre/post training assessments, and outreach metrics.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Black/African American, Latinx, or Choctaw
* Age between 18-75

Exclusion Criteria:

* Cognitive impairment
* Pregnant or plans to become pregnant within 12 months
* Currently enrolled in a food box delivery program or nutrition education program
* Food allergies that will be exacerbated with food box distribution

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-05-17 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Dietary Consumption | Baseline until 6-months following the completion of the intervention
  Visually Enhanced Food Behavior Checklist and Community Engagement Alliance (CEAL) Common Survey Questions 13-17.
  The surveys will be analyzed using a "sum of boxes" approach. Each participant has a potential score of 0-20, with higher scores indicating better dietary habits.

SECONDARY OUTCOMES:
Perceptions and Knowledge | Baseline until 6 months following the completion of the intervention
  Supplemental Nutrition Assistance Program Education (SNAP-Ed) Around the Table Survey
Dietary Intake | Baseline until 6 months following the completion of the intervention
  Automated, Self-Administered 24-hour Dietary Assessment Tool
Recruitment | Baseline until end of recruitment period
  Program registration
Retention | Baseline until completion of intervention
  Attendance log
Delivery of Intervention | Baseline until 6-months after the completion of the intervention
  Supplemental Nutrition Assistance Program Education (SNAP-Ed) Pre/Post Survey
Blood Pressure | Baseline until 6 months following the completion of the intervention
  Systolic and diastolic blood pressure, measured by study personnel using ambulatory blood pressure monitor and following AMA Cardiovascular Disease Prevention Guidelines
Blood Sugar | Baseline until 6 months following completion of the intervention
  Blood glucose levels, measured by study personnel using finger stick method
Cholesterol | Baseline until 6 months following completion of the intervention
  Lipid levels, measured by study personnel using a mobile cholesterol monitor

CONTACTS AND LOCATIONS:
Overall Officials: Caroline E Compretta, Principal Investigator — University of Mississippi Medical Center
Locations (4):
- United States (4):
  - Grace Episcopal Church, Canton, Mississippi
  - Choctaw Health Center, Choctaw, Mississippi
  - Locust Grove MB Church, Greenwood, Mississippi
  - Cade Chapel - Center for Family Life, Inc., Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with the study sponsor as outlined in Notice of Award. The study sponsor will create a database for researchers to access deidentified data across all funded sites.
Time Frame: January 2026
Access Criteria: Researchers will be able to access deidentified data from all partner sites via the NIH CEAL website.